CLINICAL TRIAL: NCT00228163
Title: Extension of Protocol HMR1726D/2001, A Phase II Study of the Safety and Efficacy of Teriflunomide (HMR1726) in Multiple Sclerosis With Relapses
Brief Title: Long Term Safety and Efficacy of Teriflunomide (HMR1726) in Multiple Sclerosis With Relapses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LTS6048; HMR1726D/2002
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis Relapsing Remitting; Secondary Progressive; Progressive Relapsing
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — teriflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teriflunomide 7 mg (Experimental)
  Interventions: Drug: teriflunomide (HMR1726)
- Teriflunomide 14 mg (Experimental)
  Interventions: Drug: teriflunomide (HMR1726)

INTERVENTIONS:
Drug: teriflunomide (HMR1726) — tablet, oral administration once daily.

SUMMARY:
The primary objective is to assess the long-term safety of teriflunomide in multiple sclerosis subjects. The secondary objective is to assess the long-term efficacy.

DETAILED DESCRIPTION:
Subjects completing the HMR 1726D/2001 study are given the opportunity to continue or switch to teriflunomide for 528 weeks or until teriflunomide is commercially available in the country where patient lives;

* subjects on Teriflunomide 7 mg or 14 mg continue on the same dose of teriflunomide.
* subjects on placebo are randomized to teriflunomide 7 mg or 14 mg.

The total study period per subject is 532 weeks or until teriflunomide is commercially available in the country where patient lives, broken up as follows:

* Treatment: 528 weeks or until teriflunomide is commercially available in the country where patient lives,
* Post-washout follow-up: 4 weeks after last treatment intake.

ELIGIBILITY:
Inclusion Criteria:

* Satisfactorily completion of HMR1726D/2001 study with respect to safety.
* If female subject, non-childbearing potential or child bearing potential with adequate contraception.
* Consent to practice/maintain adequate means of contraception throughout the study and for 24 months after the discontinuation of treatment.
* Clinically definite Multiple Sclerosis (MS) as established on entry into HMR1726D/2001 study.
* Extended Disability Status Score(EDSS) between 0 and 6 inclusively, when the subject entered HMR1726D/2001 study.
* Magnetic Resonance Imaging (MRI) criteria must continue to support the diagnosis of clinically definite MS.
* Willingness to participate in a long-term safety and efficacy trial.

Exclusion Criteria:

* Subject who did not complete HMR 1726D/2001 study for safety reasons.
* Subject who developed clinically relevant cardiovascular, hepatic, endocrine or other major disease.
* Pregnancy.
* Breast-feeding.
* Wish to parent.
* Likelihood of requiring treatment during the study period with drugs not permitted.
* Disallowed therapies such asw immunomodulators, immunosuppressants.
* Recent history of drug or alcohol abuse.
* Liver function impairment.
* Abnormal mental conditions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2002-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | Up to a maximum of 532 weeks (4 weeks after last treatment intake) or until teriflunomide is commercially available in the country where patient lives

SECONDARY OUTCOMES:
Annualized relapse rate (number of relapses per patient-year) | 528 weeks or until teriflunomide is commercially available in the country where patient lives
Change from baseline in Kurtzke Expanded Disability Status Scale (EDSS) score | 528 weeks or until teriflunomide is commercially available in the country where patient lives
Change from baseline in Multiple Sclerosis Functional Composite (MSFC) score | 528 weeks or until teriflunomide is commercially available in the country where patient lives
Burden of disease : Change from baseline in the volume of abnormal brain tissue as measured by brain Magnetic Resonance Image (MRI) | 528 weeks or until teriflunomide is commercially available in the country where patient lives
Change from baseline in Multiple Sclerosis Quality of Life Questionnaire-54 (MSQoL-54) score | 528 weeks or until teriflunomide is commercially available in the country where patient lives
Change from baseline in subject reported fatigue as assessed by the Fatigue Impact Scale (FIS) | 528 weeks or until teriflunomide is commercially available in the country where patient lives

CONTACTS AND LOCATIONS:
Overall Officials: Paul W O'Connor, MD, Principal Investigator — St. Michael's Hospital, 30 Bond Street, 3rd floor, Toronto, ON M5B 1W8, Canada
Locations (16):
- Canada (10):
  - Investigational Site Number 16, Calgary
  - Investigational Site Number 10, Halifax
  - Investigational Site Number 15, London
  - Investigational Site Number 12, Montreal
  - Investigational Site Number 11, Montreal
  - Investigational Site Number 13, Ottawa
  - Investigational Site Number 18, Québec
  - Investigational Site Number 14, Toronto
  - Investigational Site Number 17, Vancouver
  - Investigational Site Number 19, Winnipeg
- France (6):
  - Investigational Site Number 24, Clermont-Ferrand
  - Investigational Site Number 21, Lyon
  - Investigational Site Number 30, Marseille
  - Investigational Site Number 23, Montpellier
  - Investigational Site Number 28, Nice
  - Investigational Site Number 27, Rennes

REFERENCES:
- [Derived] Comi G, Freedman MS, Meca-Lallana JE, Vermersch P, Kim BJ, Parajeles A, Edwards KR, Gold R, Korideck H, Chavin J, Poole EM, Coyle PK. Prior treatment status: impact on the efficacy and safety of teriflunomide in multiple sclerosis. BMC Neurol. 2020 Oct 6;20(1):364. doi: 10.1186/s12883-020-01937-4. PMID 33023488
- [Derived] Confavreux C, Li DK, Freedman MS, Truffinet P, Benzerdjeb H, Wang D, Bar-Or A, Traboulsee AL, Reiman LE, O'Connor PW; Teriflunomide Multiple Sclerosis Trial Group. Long-term follow-up of a phase 2 study of oral teriflunomide in relapsing multiple sclerosis: safety and efficacy results up to 8.5 years. Mult Scler. 2012 Sep;18(9):1278-89. doi: 10.1177/1352458512436594. Epub 2012 Feb 3. PMID 22307384